CLINICAL TRIAL: NCT07060755
Title: Effect of Foot Bath With Peppermint Oil on Postpartum Insomnia and Fatigue Compared to Foot Bath With Warm Water Alone in the Postpartum Period
Brief Title: Effect of Different Foot Baths on Postpartum Insomnia and Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Elif Balkan, Research Assistant, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EBSOYalova
Record Dates: First submitted 2025-06-21; First posted 2025-07-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Postpartum
Keywords: fatigue; insomnia; sleepiness; footbath
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders; Sleepiness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peppermint Oil Bath Group (Experimental): This arm will have peppermint oiled footbath
  Interventions: Other: Peppermint oil footbath
- Warm water Bath Group (Experimental): This arm will have warm water footbath
  Interventions: Other: Warm Water Footbath
- Control (No Intervention): This arm will have no intervention

INTERVENTIONS:
Other: Peppermint oil footbath — This includes a footbath with peppermint oil for 30 minutes each day for 2 weeks
  Arms: Peppermint Oil Bath Group
Other: Warm Water Footbath — This includes a warm water footbath for 30 minutes each day dor 2 weeks
  Arms: Warm water Bath Group

SUMMARY:
The goal of this clinical trial is to assess if different footbaths works to decrease postpartum fatigue and insomnia. The main questions are:

Does peppermint oil footbaths decrease fatigue and insomnia in postpartum period? Does peppermint oil footbaths more effective than footbaths with warm water?

Researchers will compare peppermint oil footbath, warm water footbath to no intervention.

Participants will:

Answer some scales and questionnaire. Do peppermint oil footbath or warm water footbath for 30 minutes each day postpartum during 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Giving birth at term (38-42 weeks of gestation)
* Being within the first 24 hours postpartum
* Participating in the study voluntarily
* Being over 18 years of age

Exclusion Criteria:

* Having a risky pregnancy diagnosis
* Having complications during and after birth
* Having a cardiovascular system disease diagnosis
* Having an open wound in the foot area
* Having any skin problems in the foot area (such as fungus)
* Having communication problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender people identify with the gender that aligns with the sex they were assigned at birth
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 1st day to the 14th day
  Fatigue will be assessed via Postnatal Accumulated Fatigue Scale. This scale used to assess the fatigue levels of postpartum women in the postpartum period. The scale consists of a total of 13 items and 3 sub-dimensions answered as "almost none," "sometimes," and "mostly." The items of the scale are scored between 0 and 3, and as the total score increases, it is interpreted that the individual's fatigue increases. The scale has no cut-off score.
Postpartum Sleep Quality | 1st day to 14th day
  Postpartum Sleep Quality Scale will use to assess sleep quality. This scale aims to evaluate sleep quality in the postpartum period. The scale has a 5-point Likert structure and consists of a total of 14 items and three sub-dimensions. Scale items are scored between 0 and 4. The score that can be obtained from the scale varies between 0-56.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly due to ethical restrictions. But authors may share IPD with researchers who reach out to the authors for data sharing with necessary reasons

REFERENCES:
- [Background] Kirca AS, Gul DK, Sener N. Psychometric properties of postnatal accumulated fatigue scale validity and reliability. J Obstet Gynaecol Res. 2023 Jul;49(7):1762-1769. doi: 10.1111/jog.15651. Epub 2023 Apr 23. PMID 37088932